CLINICAL TRIAL: NCT03720470
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER STUDY INVESTIGATING THE EFFICACY AND SAFETY OF PF-04965842 AND DUPILUMAB IN COMPARISON WITH PLACEBO IN ADULT SUBJECTS ON BACKGROUND TOPICAL THERAPY, WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study Evaluating Efficacy and Safety of PF-04965842 and Dupilumab in Adult Subjects With Moderate to Severe Atopic Dermatitis on Background Topical Therapy
Acronym: JADE Compare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451029; COMPARE (Other: Alias Study Number); 2018-002573-21 (EudraCT Number)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Dermatitis; Dermatitis, Atopic; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases | interventions — abrocitinib; dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PF-04965842 100 mg + Placebo Inj followed by PF-04965842 100mg (Experimental): Once-daily oral PF-04965842 100 mg + Placebo injected subcutaneously once every 2 weeks from Day 1 until Week 16 followed by once-daily oral PF-04965842 100 mg from Week 16 to Week 20
  Interventions: Drug: PF-04965842 100 mg; Drug: Injectable Placebo
- PF-04965842 200 mg + Placebo Inj followed by PF-04965842 200mg (Experimental): Once-daily oral PF-04965842 200 mg + Placebo injected subcutaneously once every 2 weeks from Day 1 until Week 16 followed by once-daily oral PF-04965842 200 mg from Week 16 to Week 20
  Interventions: Drug: PF-04965842 200 mg; Drug: Injectable Placebo
- Dupilumab Injection + Oral Placebo followed by Oral Placebo (Active Comparator): Dupilumab injected subcutaneously once every 2 weeks + once-daily oral Placebo from Day 1 until Week 16 followed by once-daily oral Placebo from Week 16 to Week 20
  Interventions: Drug: Dupilumab; Drug: Oral Placebo
- Oral Placebo + Placebo Inj followed by 100 mg PF-04965842 (Placebo Comparator): Once-daily oral Placebo + Placebo injected subcutaneously once every 2 weeks from Day 1 until Week 16 followed by once-daily oral 100 mg PF-04965842 from Week 16 to Week 20
  Interventions: Drug: PF-04965842 100 mg; Drug: Oral Placebo; Drug: Injectable Placebo
- Oral Placebo + Placebo Inj followed by 200 mg PF-04965842 (Placebo Comparator): Once-daily oral Placebo + Placebo injected subcutaneously once every 2 weeks from Day 1 until Week 16 followed by once-daily oral 200 mg PF-04965842 from Week 16 to Week 20
  Interventions: Drug: PF-04965842 200 mg; Drug: Oral Placebo; Drug: Injectable Placebo

INTERVENTIONS:
Drug: PF-04965842 100 mg — PF-04965842 100 mg, administered as two tablets to be taken orally once daily as follows:
  1. In the arm "PF-04965842 100 mg + Injectable Placebo followed by PF-04965842 100 mg," PF-04965842 100 mg is taken together with Injectable Placebo from Day 1 until Week 16, then by itself from Week 16 to Week 20;
  2. In the arm "Oral Placebo + Injectable Placebo followed by 100 mg PF-04965842" subjects take PF-04965842 100 mg from Week 16 to Week 20.
  Arms: Oral Placebo + Placebo Inj followed by 100 mg PF-04965842; PF-04965842 100 mg + Placebo Inj followed by PF-04965842 100mg
Drug: PF-04965842 200 mg — PF-04965842 200 mg, administered as two tablets to be taken orally once daily as follows:
  1. In the arm "PF-04965842 200 mg + Injectable Placebo followed by PF-04965842 100 mg," PF-04965842 200 mg is taken together with Injectable Placebo from Day 1 until Week 16, then by itself from Week 16 to Week 20;
  2. In the arm "Oral Placebo + Injectable Placebo followed by 200 mg PF-04965842" subjects take PF-04965842 200 mg from Week 16 to Week 20.
  Arms: Oral Placebo + Placebo Inj followed by 200 mg PF-04965842; PF-04965842 200 mg + Placebo Inj followed by PF-04965842 200mg
Drug: Dupilumab — Two subcutaneous injections of Dupilumab 300 mg as a loading dose administered on Day 1 (for a total of 600 mg) followed by one injection once every two weeks (q2w) until Week 16.
  Arms: Dupilumab Injection + Oral Placebo followed by Oral Placebo
Drug: Oral Placebo — Oral placebo (for PF-04965842) administered as two tablets to be taken orally once daily as follows:
  1. In the arm "Dupilumab Injection + Oral Placebo followed by Oral Placebo," the Oral Placebo is taken together with Dupilumab from Day 1 until Week 16, then by itself to Week 20;
  2. In the arms "Oral Placebo + Injectable Placebo followed by 100 mg PF-04965842" and "Oral Placebo + Injectable Placebo followed by 200 mg PF-04965842," subjects, take Oral Placebo from Day 1 until Week 16.
  Arms: Dupilumab Injection + Oral Placebo followed by Oral Placebo; Oral Placebo + Placebo Inj followed by 100 mg PF-04965842; Oral Placebo + Placebo Inj followed by 200 mg PF-04965842
Drug: Injectable Placebo — Two subcutaneous injections of Placebo (for Dupilumab) administered as a loading dose on Day 1 followed by one injection every other week (q2w) until Week 16.
  Arms: Oral Placebo + Placebo Inj followed by 100 mg PF-04965842; Oral Placebo + Placebo Inj followed by 200 mg PF-04965842; PF-04965842 100 mg + Placebo Inj followed by PF-04965842 100mg; PF-04965842 200 mg + Placebo Inj followed by PF-04965842 200mg

SUMMARY:
B7451029 is a Phase 3 study to investigate PF-04965842 in adult patients who have moderate to severe atopic dermatitis and use background topical therapy. The efficacy of two dosage strengths of PF-04965842, 100 mg and 200 mg taken orally once daily will be evaluated relative to placebo over 12 weeks. The efficacy of the two dosage strengths of PF-04965842 will be compared with dupilumab in terms of pruritus relief at 2 weeks. The two dosage strengths of PF-04965842 and dupilumab 300 mg injected subcutaneously once every two weeks (with a loading dose of 600 mg injected on the first day) will also be evaluated relative to placebo over 16 weeks. The safety of the investigational products will be evaluated over the duration of the study. Subjects will use non-medicated emollient at least twice a day and medicated topical therapy such as corticosteroids, calcineurin inhibitors or PDE4 inhibitors, as per protocol guidance, to treat active lesions during the study. Subjects who are randomized to receive one of the two dosage strengths of PF-04965842 will also receive placebo injectable study drug every two weeks until Week 16 and then will continue on receiving only the oral study drug for 4 weeks. Subjects who are randomized to receive dupilumab injections every two weeks will also receive oral placebo to be taken once daily until Week 16 and will then continue to receive only the oral placebo for 4 weeks. Subjects who are randomized to the placebo arms, will receive both daily oral placebo and injectable placebo every two weeks until Week 16, after which they will receive either 100 mg or 200 mg of PF-04965842 taken orally once daily for 4 weeks, dependent upon which arm they have been allocated to. Eligible subjects will have an option to enter a long-term extension study after completing 20 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older at the time of informed consent
* Diagnosis of atopic dermatitis (AD) for at least 1 year and current status of moderate to severe disease (>= the following scores: BSA 10%, IGA 3, EASI 16, Pruritus NRS severity 4)
* Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with medicated topical therapy for AD for at least 4 weeks, or who have required systemic therapies for control of their disease.
* Must be willing and able to comply with standardized background topical therapy, as per protocol guidelines throughout the study
* Female subjects who are of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

  1. Female subjects of childbearing potential must have a confirmed negative pregnancy test prior to randomization;
  2. Female subjects of childbearing potential must agree to use a highly effective method of contraception for the duration of the active treatment period and for at least 28 days after the last dose of investigational product.
* Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  * Have medically confirmed ovarian failure; or
  * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state.

All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.

-If receiving concomitant medications for any reason other than AD, must be on a stable regimen prior to Day 1 and through the duration of the study

Exclusion Criteria:

* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Other active nonAD inflammatory skin diseases or conditions affecting skin
* Prior treatment with JAK inhibitors
* Previous treatment with dupilumab
* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (215):
- United States (60):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - The University Of Alabama At Birmingham, Birmingham, Alabama
  - Marvel Research, LLC, Huntington Beach, California
  - Alliance Research Centers, Laguna Hills, California
  - Allergy & Asthma Care Center of Southern California, Long Beach, California
  - Allergy & Asthma Associates of Southern California dba Southern California Research, Mission Viejo, California
  - Dermatology Specialists, Inc., Murrieta, California
  - MedDerm Associates, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Synexus Clinical Research US, Inc., Santa Rosa, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Renaissance Research and Medical Group, Inc, Cape Coral, Florida
  - C & R Research Services USA, Inc, Coral Gables, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Olympian Clinical Research, Largo, Florida
  - Savin Medical Group LLC, Miami, Florida
  - Wellness Clinical Research, LLC, Miami Lakes, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Research Institute of Southeast, LLC, West Palm Beach, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Idaho Allergy and Research, Eagle, Idaho
  - ASR, LLC, Nampa, Idaho
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Midwest Allergy Sinus Asthma, SC, Normal, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Forefront Dermatology, S.C., Louisville, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Skin Laser and Surgery Specialists of NY and NJ, Hackensack, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Juva Skin and Laser Center, New York, New York
  - TrialSpark, Inc (Russell Cohen), Oceanside, New York
  - Cary Dermatology Center, PA, Cary, North Carolina
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research Inc., d/b/a PMG Research of Piedmont HealthCare, Statesville, North Carolina
  - Winston-Salem Dermatology and Surgery Center, PLLC, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Portland Clinical Research dba Columbia Allergy & Asthma Clinic, Clackamas, Oregon
  - Crisor, LLC, Medford, Oregon
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Synexus Clinical Research US. Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Arlington Research Center, Inc., Arlington, Texas
  - Austin Institute for Clinical Research, Inc., Austin, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
  - Velocity Urgent Care, Norfolk, Virginia
- Australia (10):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Australian Clinical Research Network, Maroubra, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - North Eastern Health Specialists, Hectorville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Skin and Cancer Foundation Inc, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (6):
  - DCC 2/Sofia EOOD, Sofia
  - "DCC Aleksandrovska" EOOD, Sofia
  - Dermatology Clinic "Sofia" Ltd, Sofia
  - "Mc Synexus Sofia" Eood, Sofia
  - Medical Centre Synexus Sofia EOOD-branch Stara Zagora, Stara Zagora
  - "DCC "Mladost-M Varna" OOD, Varna
- Canada (11):
  - Pacific Dermaesthetics Inc., Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - AvantDerm Clinical Research, Toronto, Ontario
  - Manna Research (Toronto), Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Dr. Rachel Asiniwasis Medical Prof Corp, Regina, Saskatchewan
- Chile (4):
  - Centro Medico SkinMed Limitada, Santiago, Santiago Metropolitan
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
  - MIRES (M y F Estudios Clínicos Limitada), Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
- Czechia (9):
  - Dermamedica S.R.O., Náchod
  - CCR Ostrava, s.r.o., Ostrava
  - BENU Lekarna, Pardubice
  - CCR Czech, a.s., Pardubice
  - Nemocnice Pardubickeho kraje a.s., Pardubicka nemocnice, odd Dermatologie, Pardubice
  - Sanatorium profesora Arenbergera, Prague
  - Lekarna U sv. Ignace, Prague
  - Synexus Czech, s.r.o., Prague
  - CCR Prague, s.r.o., Prague
- Germany (15):
  - Licca Clinical Research Institute, Augsburg
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Klinikum Bielefeld Rosenhohe, Bielefeld
  - Universitätsklinikum Bonn AöR, Bonn
  - Klinische Forschung Dresden GmbH, Dresden
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - IKF Pneumologie GmbH & Co KG, Institut fuer klinische Forschung, Frankfurt
  - Universitätsklinikum und Poliklinik für Dermatologie und Venerologie, Halle
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Studienzentrum Dr. med. Beate Schwarz, Langenau
  - SIBAmed Studienzentrum GmbH & Co KG, Leipzig
  - Universitaetsklinikum Schleswig-Holstein/Campus Luebeck, Lübeck
  - Dermatologische Gemeinschaftspraxis Dres. Scholz, Sebastian, Schilling, Mahlow
  - Universitätsklinikum Marburg, Marburg
  - University of Muenster, Münster
- Hungary (5):
  - SE AOK Bor-, Nemikortani es Boronkologiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. Synexus Gyula DRS, Gyula
  - Trial Pharma Kft., Püspökladány
  - Medmare Bt, Veszprém
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS Universita Cattolica del Sacro Cuore, Roma, RM
  - AOU Policlinico di Modena, Struttura Complessa di Dermatologia, Modena
- Japan (12):
  - Kawashima Dermatology Clinic, Ichikawa, Chiba
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Dermatology Shimizu Clinic, Kobe, Hyōgo
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Kume Clinic, Sakai, Osaka
  - Iidabashi Skin Clinic, Chiyoda-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjyuku-ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
  - Sanrui Hifuka, Saitama
- Latvia (5):
  - Riga 1st Hospital, Clinic for Dermatology and STD, Riga
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Childrens Clinical University Hospital State SLLC, Riga
  - Health and aesthetics Ltd, Riga
  - Outpatient Clinic of Ventspils, Ventspils
- Mexico (4):
  - Cryptex Investigación Clínica, S.A. de C.V., Cuauhtémoc, Mexico City
  - Arke Estudios Clinicos S.A. de C.V., Cuauhtémoc, Mexico City
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - SMIQ. S. de R. L. de C.V., Querétaro
- Poland (38):
  - NZOZ Specjalistyczny Osrodek Dermatologiczny "DERMAL", Bialystok
  - Centrum Medyczne SENSEMED, Chorzów
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - COPERNICUS-SZPITAL Oddzial Dermatologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Dermatologii, Wenerologii i Alergologii, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - MCBK, Grodzisk Mazowiecki
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Care Clinic Centrum Medyczne, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Gabinet Dermatologiczny Beata Krecisz, Kielce
  - Centrum Medyczne Plejady, Krakow
  - AWP Klinika Dermatologii Pod Fortem Anna Wojas-Pelc, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Medyczne Promed, Krakow
  - Prywatna Praktyka Lekarska - Adam Smialowski, Ksawerów
  - Dermoklinika-Centrum Medyczne s.c. M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Salve Medica Sp. z o.o. Sp. k., Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - NZOZ "Med-Laser" Borzecki Spolka Jawna, Lublin
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan
  - Clinical Research Center Spolka z ograniczona odpowiedzialnoscia MEDIC-R Sp.k., Poznan
  - LIFT-MED Spolka Akcyjna, Rybnik
  - Kliniczny Szpital Wojewodzki nr 1 im. F. Chopina, Klinika Dermatologii, Rzeszów
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Medycyna Kliniczna, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - RCMed Oddzial Warszawa, Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - "REUMATIKA - Centrum Reumatologii" NZOZ, Warsaw
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej, Wroclaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Lukasz Matusiak "4Health", Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Slovakia (5):
  - SUMMIT CLINICAL RESEARCH, s.r.o., Bratislava
  - Nemocnica Kosice-Saca, a.s., 1. sukromna nemocnica, Kosice-Saca
  - Pedi-Derma s.r.o., Košice
  - Fakultna nemocnica s poliklinikou Nove Zamky, Dermatovenerologicka Klinika, Nové Zámky
  - SANARE spol. s.r.o., Dermatovenerologicka ambulancia, Svidník
- South Korea (7):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Chungnam National University Hospital CNUH, Daejeon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Yonsei Univ. Health System, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (6):
  - Taipei Veterans General Hospital, Taipei, Taiwan (r.o.c)
  - Chung Shan Medical University Hospital (CSMUH), Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- United Kingdom (11):
  - Medinova Research -West London Dedicated Research Centre, Wokingham, Berkshire
  - Derriford Hospital, Plymouth, Devon
  - Medinova Research, East London Dedicated Research Centre, Romford, Essex
  - Guy's Hospital-Guy's and St Thomas NHS Foundation Trust, London, Greater London
  - Medinova Research, South London Clinical Trial Centre, Sidcup, KENT
  - MeDiNova Research North London Dedicated Research Centre, Northwood, Middlesex
  - Medinova Research, Yaxley, Peterborough
  - Medinova Research, Warwickshire Dedicated Research Centre, Kenilworth, Warwickshire
  - Medinova, Yorkshire Quality Research Site, Shipley, WEST Yorkshire
  - MeDiNova Northamptonshire Dedicated Research Centre, Corby
  - West Glasgow ACH, NHS Greater Glasgow and Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Simpson EL, Silverberg JI, Geng B, Carrascosa JM, Bieber T, Brunner PM, Staumont-Salle D, Ji C, Biswas P, Feeney C, Hernandez-Martin I, Rebollo Laserna FJ, Koppensteiner H. Do Allergic Comorbidities Alter the Efficacy and Safety of Abrocitinib or Dupilumab in Patients with Moderate-to-Severe Atopic Dermatitis? Dermatol Ther (Heidelb). 2025 Nov;15(11):3391-3407. doi: 10.1007/s13555-025-01516-w. Epub 2025 Sep 23. PMID 40987931
- [Derived] Silverberg JI, Thyssen JP, Lazariciu I, Myers DE, Guler E, Chovatiya R. Abrocitinib may improve itch and quality of life in patients with itch-dominant atopic dermatitis. Skin Health Dis. 2024 May 5;4(4):e382. doi: 10.1002/ski2.382. eCollection 2024 Aug. PMID 39104653
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Simpson EL, Silverberg JI, Thyssen JP, Viguier M, Thaci D, de Bruin-Weller M, Weidinger S, Chan G, DiBonaventura M, Biswas P, Feeney C, Koulias C, Cork MJ. Efficacy and Safety of Abrocitinib in Patients with Severe and/or Difficult-to-Treat Atopic Dermatitis: A Post Hoc Analysis of the Randomized Phase 3 JADE COMPARE Trial. Am J Clin Dermatol. 2023 Jul;24(4):609-621. doi: 10.1007/s40257-023-00785-5. Epub 2023 May 22. PMID 37213005
- [Derived] Stander S, Kwatra SG, Silverberg JI, Simpson EL, Thyssen JP, Yosipovitch G, Zhang F, Cameron MC, Cella RR, Valdez H, DiBonaventura M, Feeney C. Early Itch Response with Abrocitinib Is Associated with Later Efficacy Outcomes in Patients with Moderate-to-Severe Atopic Dermatitis: Subgroup Analysis of the Randomized Phase III JADE COMPARE Trial. Am J Clin Dermatol. 2023 Jan;24(1):97-107. doi: 10.1007/s40257-022-00738-4. Epub 2022 Dec 13. PMID 36512175
- [Derived] Reich K, Lio PA, Bissonnette R, Alexis AF, Lebwohl MG, Pink AE, Kabashima K, Boguniewicz M, Nowicki RJ, Valdez H, Zhang F, DiBonaventura M, Cameron MC, Clibborn C. Magnitude and Time Course of Response to Abrocitinib for Moderate-to-Severe Atopic Dermatitis. J Allergy Clin Immunol Pract. 2022 Dec;10(12):3228-3237.e2. doi: 10.1016/j.jaip.2022.08.042. Epub 2022 Sep 13. PMID 36108923
- [Derived] Alexis A, de Bruin-Weller M, Weidinger S, Soong W, Barbarot S, Ionita I, Zhang F, Valdez H, Clibborn C, Yin N. Rapidity of Improvement in Signs/Symptoms of Moderate-to-Severe Atopic Dermatitis by Body Region with Abrocitinib in the Phase 3 JADE COMPARE Study. Dermatol Ther (Heidelb). 2022 Mar;12(3):771-785. doi: 10.1007/s13555-022-00694-1. Epub 2022 Mar 17. PMID 35297025
- [Derived] Bieber T, Simpson EL, Silverberg JI, Thaci D, Paul C, Pink AE, Kataoka Y, Chu CY, DiBonaventura M, Rojo R, Antinew J, Ionita I, Sinclair R, Forman S, Zdybski J, Biswas P, Malhotra B, Zhang F, Valdez H. Comparing abrocitinib and dupilumab in the treatment of atopic dermatitis: a plain language summary. Immunotherapy. 2022 Jan;14(1):5-14. doi: 10.2217/imt-2021-0224. Epub 2021 Nov 15. PMID 34775830
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- [Derived] Bieber T, Simpson EL, Silverberg JI, Thaci D, Paul C, Pink AE, Kataoka Y, Chu CY, DiBonaventura M, Rojo R, Antinew J, Ionita I, Sinclair R, Forman S, Zdybski J, Biswas P, Malhotra B, Zhang F, Valdez H; JADE COMPARE Investigators. Abrocitinib versus Placebo or Dupilumab for Atopic Dermatitis. N Engl J Med. 2021 Mar 25;384(12):1101-1112. doi: 10.1056/NEJMoa2019380. PMID 33761207
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had treatment period of 20 weeks. The first part of this treatment period consists of a 16-week randomized, double-blind, placebo-controlled, double-dummy treatment period where participants received PF-04965842, dupilumab and placebo. The randomization and double-blind was maintained during the final 4 weeks of the treatment period, but participants only received PF-04965842 and placebo.
Groups:
- Placebo up to Week 16: Participants were randomized to receive oral placebo matched to PF-04965842 once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 till Week 16.
- Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20: Participants who were randomized to receive oral placebo matched to PF-04965842 with subcutaneous injectable placebo matched to dupilumab till Week 16, received PF-04965842 100 milligram (mg) tablet orally once daily post Week 16 up to Week 20.
- Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20: Participants who were randomized to receive oral placebo matched to PF-04965842 with subcutaneous injectable placebo matched to dupilumab till Week 16, received PF-04965842 200 mg tablet orally once daily post Week 16 up to Week 20.
- PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20: Participants were randomized to receive PF-04965842 100 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16, followed by administration of PF-04965842 100 mg tablet orally once daily post Week 16 up to Week 20.
- PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20: Participants were randomized to receive PF-04965842 200 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16, followed by administration of PF-04965842 200 mg tablet orally once daily post Week 16 up to Week 20.
- Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20: Participants were randomized to receive dupilumab 300 mg subcutaneous injection every other week with oral placebo matched to PF-04965842 once daily from Day 1 to Week 16, followed by administration of oral placebo matched to PF-04965842 once daily post Week 16 up to Week 20.
Period: Treatment Period: First Part 16 Weeks
Arm/Group | Placebo up to Week 16 | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Started | 131 | 0 | 0 | 238 | 226 | 243
Treated/ Safety Analysis Set | 131 | 0 | 0 | 238 | 226 | 242
Full Analysis Set | 131 | 0 | 0 | 238 | 226 | 242
Completed | 117 | 0 | 0 | 217 | 208 | 223
Not Completed | 14 | 0 | 0 | 21 | 18 | 20
Not completed — Adverse Event | 5 | 0 | 0 | 5 | 8 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol deviation | 2 | 0 | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 9 | 3 | 6
Not completed — Medication Error Without Associated Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 1 | 2 | 2
Not completed — Randomized But Not Treated | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period: Final 4 Weeks
Arm/Group | Placebo up to Week 16 | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Started | 0 (Participants received placebo till Week 16 then allocated to receive PF-04965842 post Week 16.) | 60 (Participants received placebo till Week 16 then allocated to receive PF-04965842 post Week 16.) | 57 (Participants received placebo till Week 16 then allocated to receive PF-04965842 post Week 16.) | 217 | 208 | 223
Treated/ Safety Analysis Set | 0 | 60 | 57 | 217 | 208 | 223
Full Analysis Set | 0 | 60 | 57 | 217 | 208 | 223
Completed | 0 | 58 | 55 | 210 | 204 | 218
Not Completed | 0 | 2 | 2 | 7 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 2 | 2
Not completed — Other | 0 | 1 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20 | Total
Number analyzed (Participants) | 131 | 238 | 226 | 242 | 837
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 121 | 224 | 211 | 227 | 783
  >=65 years | 10 | 14 | 15 | 15 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 118 | 122 | 134 | 428
  Male | 77 | 120 | 104 | 108 | 409
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 35 | 36 | 37 | 124
  Not Hispanic or Latino | 113 | 200 | 187 | 201 | 701
  Unknown or Not Reported | 2 | 3 | 3 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 2 | 5
  Asian | 31 | 48 | 53 | 46 | 178
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 6 | 6 | 9 | 14 | 35
  White | 87 | 182 | 161 | 176 | 606
  More than one race | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 3 | 0 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) or Almost Clear (1) and a Reduction of Greater Than or Equal to (>=) 2 Points From Baseline at Week 12
Description: IGA assessed severity of atopic dermatitis (AD) on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded scalp, palms and sole.
Time Frame: Baseline (the last measurement prior to first dosing on Day 1), Week 12
Population: Full analysis set till Week 16 included all randomized participants who received at least 1 dose of study medication up to Week 16. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PF-04965842 100 mg + Placebo Injection up to Week 16: Participants were randomized to receive PF-04965842 100 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16.
- PF-04965842 200 mg + Placebo Injection up to Week 16: Participants were randomized to receive PF-04965842 200 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16.
- Dupilumab 300 mg + Oral Placebo up to Week 16: Participants were randomized to receive dupilumab 300 mg subcutaneous injection every other week with oral placebo matched to PF-04965842 once daily from Day 1 to Week 16.
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 129 | 235 | 219 | 241
Percentage of participants | 14.0 [8.0 to 19.9] | 36.6 [30.4 to 42.8] | 48.4 [41.8 to 55.0] | 36.5 [30.4 to 42.6]
Statistical Analysis 1: Comparison: Placebo up to Week 16 vs PF-04965842 100 mg + Placebo Injection up to Week 16; Difference in percentage (PF-04965842 versus placebo) and confidence interval (CI) for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 23.1, 95% CI 2-sided [14.7 to 31.4]
Statistical Analysis 2: Comparison: Placebo up to Week 16 vs PF-04965842 200 mg + Placebo Injection up to Week 16; Difference in percentage (PF-04965842 versus placebo) and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 34.8, 95% CI 2-sided [26.1 to 43.5]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >=75 Percent (%) Improvement From Baseline at Week 12
Description: EASI evaluates severity of participants with AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 129 | 235 | 219 | 241
Percentage of participants | 27.1 [19.5 to 34.8] | 58.7 [52.4 to 65.0] | 70.3 [64.3 to 76.4] | 58.1 [51.9 to 64.3]
Statistical Analysis 1: Comparison: Placebo up to Week 16 vs PF-04965842 100 mg + Placebo Injection up to Week 16; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 31.9, 95% CI 2-sided [22.2 to 41.6]
Statistical Analysis 2: Comparison: Placebo up to Week 16 vs PF-04965842 200 mg + Placebo Injection up to Week 16; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 43.2, 95% CI 2-sided [33.7 to 52.7]

3. Secondary Outcome: Percentage of Participants With at Least 4 Points Improvement in the Numerical Rating Scale (NRS) for Severity of Pruritus From Baseline at Day 2-15, Week 2, 4, 8, 12 and 16
Description: Participants were asked to assess their worst pruritus/itching due to AD over the past 24 hours on an NRS scale ranged from 0 (no itching) to 10 (worst possible itching), where higher scores indicated greater severity.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and Week 2, 4, 8, 12, 16
Population: Full analysis set till Week 16 included all randomized participants who received at least 1 dose of study medication up to Week 16. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Day 2: number analyzed (Participants) | 117 | 220 | 203 | 206
  Day 2 | 5.1 [1.1 to 9.1] | 5.9 [2.8 to 9.0] | 7.4 [3.8 to 11.0] | 2.4 [0.3 to 4.5]
  Day 3: number analyzed (Participants) | 114 | 214 | 203 | 213
  Day 3 | 7.9 [2.9 to 12.8] | 8.4 [4.7 to 12.1] | 14.8 [9.9 to 19.7] | 3.3 [0.9 to 5.7]
  Day 4: number analyzed (Participants) | 116 | 216 | 199 | 216
  Day 4 | 6.0 [1.7 to 10.4] | 11.6 [7.3 to 15.8] | 18.6 [13.2 to 24.0] | 5.6 [2.5 to 8.6]
  Day 5: number analyzed (Participants) | 119 | 211 | 196 | 210
  Day 5 | 7.6 [2.8 to 12.3] | 14.2 [9.5 to 18.9] | 26.5 [20.3 to 32.7] | 9.5 [5.6 to 13.5]
  Day 6: number analyzed (Participants) | 119 | 213 | 207 | 214
  Day 6 | 10.9 [5.3 to 16.5] | 15.0 [10.2 to 19.8] | 25.1 [19.2 to 31.0] | 14.0 [9.4 to 18.7]
  Day 7: number analyzed (Participants) | 108 | 214 | 208 | 216
  Day 7 | 11.1 [5.2 to 17.0] | 20.1 [14.7 to 25.5] | 28.8 [22.7 to 35.0] | 13.4 [8.9 to 18.0]
  Day 8: number analyzed (Participants) | 118 | 210 | 207 | 212
  Day 8 | 14.4 [8.1 to 20.7] | 21.4 [15.9 to 27.0] | 33.3 [26.9 to 39.8] | 16.5 [11.5 to 21.5]
  Day 9: number analyzed (Participants) | 115 | 204 | 208 | 209
  Day 9 | 13.0 [6.9 to 19.2] | 24.0 [18.2 to 29.9] | 34.1 [27.7 to 40.6] | 14.8 [10.0 to 19.7]
  Day 10: number analyzed (Participants) | 114 | 203 | 207 | 210
  Day 10 | 13.2 [7.0 to 19.4] | 25.6 [19.6 to 31.6] | 34.3 [27.8 to 40.8] | 17.1 [12.0 to 22.2]
  Day 11: number analyzed (Participants) | 118 | 201 | 210 | 210
  Day 11 | 12.7 [6.7 to 18.7] | 25.4 [19.4 to 31.4] | 39.5 [32.9 to 46.1] | 20.5 [15.0 to 25.9]
  Day 12: number analyzed (Participants) | 117 | 204 | 202 | 215
  Day 12 | 12.0 [6.1 to 17.8] | 25.5 [19.5 to 31.5] | 44.1 [37.2 to 50.9] | 21.9 [16.3 to 27.4]
  Day 13: number analyzed (Participants) | 114 | 196 | 203 | 212
  Day 13 | 13.2 [7.0 to 19.4] | 30.6 [24.2 to 37.1] | 43.8 [37.0 to 50.7] | 23.6 [17.9 to 29.3]
  Day 14: number analyzed (Participants) | 121 | 210 | 199 | 212
  Day 14 | 15.7 [9.2 to 22.2] | 31.4 [25.1 to 37.7] | 45.7 [38.8 to 52.7] | 24.5 [18.7 to 30.3]
  Day 15: number analyzed (Participants) | 117 | 207 | 208 | 211
  Day 15 | 11.1 [5.4 to 16.8] | 30.4 [24.2 to 36.7] | 49.0 [42.2 to 55.8] | 26.5 [20.6 to 32.5]
  Week 2: number analyzed (Participants) | 130 | 236 | 226 | 239
  Week 2 | 13.8 [7.9 to 19.8] | 31.8 [25.8 to 37.7] | 49.1 [42.6 to 55.6] | 26.4 [20.8 to 31.9]
  Week 4: number analyzed (Participants) | 124 | 224 | 214 | 232
  Week 4 | 20.2 [13.1 to 27.2] | 44.6 [38.1 to 51.2] | 59.3 [52.8 to 65.9] | 45.3 [38.9 to 51.7]
  Week 8: number analyzed (Participants) | 122 | 221 | 214 | 229
  Week 8 | 27.0 [19.2 to 34.9] | 47.5 [40.9 to 54.1] | 64.0 [57.6 to 70.4] | 50.7 [44.2 to 57.1]
  Week 12: number analyzed (Participants) | 121 | 221 | 217 | 224
  Week 12 | 28.9 [20.8 to 37.0] | 47.5 [40.9 to 54.1] | 63.1 [56.7 to 69.6] | 54.5 [47.9 to 61.0]
  Week 16: number analyzed (Participants) | 94 | 168 | 172 | 189
  Week 16 | 28.7 [19.6 to 37.9] | 47.0 [39.5 to 54.6] | 62.8 [55.6 to 70.0] | 57.1 [50.1 to 64.2]
Statistical Analysis 1: Comparison: Placebo up to Week 16 vs PF-04965842 100 mg + Placebo Injection up to Week 16; Week 2: Difference in percentage (PF-04965842 versus placebo) and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Difference in percentage = 17.9, 95% CI 2-sided [9.5 to 26.3]
Statistical Analysis 2: Comparison: Placebo up to Week 16 vs PF-04965842 200 mg + Placebo Injection up to Week 16; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Percentage = 34.9, 95% CI 2-sided [26.0 to 43.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg + Placebo Injection up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; Week 2: Difference in percentage (PF-04965842 versus dupilumab) and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Superiority; p = 0.2084, Cochran-Mantel-Haenszel; Difference in Percentage = 5.2, 95% CI 2-sided [-2.9 to 13.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg + Placebo Injection up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 22.1, 95% CI 2-sided [13.5 to 30.7]

4. Secondary Outcome: Percentage of Participants Achieving IGA Response of Clear (0) or Almost Clear (1) and a Reduction of >=2 Points From Baseline at Week 2, 4, 8 and 16
Description: IGA assessed severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded sole, palms and scalp.
Time Frame: Baseline, Week 2, 4, 8 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 230 | 223 | 236
  Week 2 | 6.3 [2.1 to 10.4] | 15.2 [10.6 to 19.9] | 18.4 [13.3 to 23.5] | 4.7 [2.0 to 7.4]
  Week 4: number analyzed (Participants) | 129 | 234 | 223 | 238
  Week 4 | 6.2 [2.0 to 10.4] | 25.2 [19.6 to 30.8] | 31.4 [25.3 to 37.5] | 18.9 [13.9 to 23.9]
  Week 8: number analyzed (Participants) | 129 | 232 | 225 | 239
  Week 8 | 10.1 [4.9 to 15.3] | 35.8 [29.6 to 41.9] | 50.7 [44.1 to 57.2] | 28.5 [22.7 to 34.2]
  Week 16: number analyzed (Participants) | 124 | 230 | 221 | 232
  Week 16 | 12.9 [7.0 to 18.8] | 34.8 [28.6 to 40.9] | 47.5 [40.9 to 54.1] | 38.8 [32.5 to 45.1]
Statistical Analysis 1: Comparison: Placebo up to Week 16 vs PF-04965842 100 mg + Placebo Injection up to Week 16; Week 16: Difference in percentage (PF-04965842 versus placebo) and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 22.1, 95% CI 2-sided [13.7 to 30.5]
Statistical Analysis 2: Comparison: Placebo up to Week 16 vs PF-04965842 200 mg + Placebo Injection up to Week 16; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 35.0, 95% CI 2-sided [26.3 to 43.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg + Placebo Injection up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; Week 16: Difference in percentage (PF-04965842 versus dupilumab) and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions. P-value was adjusted by baseline disease severity; Test type: Other; Difference in Percentage = -3.5, 95% CI 2-sided [-12.2 to 5.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg + Placebo Injection up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; [analysis description as in outcome 4, analysis 3]; Test type: Other; Difference in Percentage = 9.4, 95% CI 2-sided [0.4 to 18.5]

5. Secondary Outcome: Percentage of Participants Achieving EASI Response >=75% Improvement From Baseline at Week 2, 4, 8 and 16
Description: EASI evaluates severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 2, 4, 8 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 228 | 223 | 235
  Week 2 | 10.9 [5.5 to 16.3] | 25.4 [19.8 to 31.1] | 30.0 [24.0 to 36.1] | 14.0 [9.6 to 18.5]
  Week 4: number analyzed (Participants) | 128 | 233 | 223 | 238
  Week 4 | 15.6 [9.3 to 21.9] | 44.6 [38.3 to 51.0] | 57.4 [50.9 to 63.9] | 38.2 [32.1 to 44.4]
  Week 8: number analyzed (Participants) | 129 | 232 | 224 | 239
  Week 8 | 18.6 [11.9 to 25.3] | 55.6 [49.2 to 62.0] | 67.9 [61.7 to 74.0] | 52.7 [46.4 to 59.0]
  Week 16: number analyzed (Participants) | 124 | 229 | 221 | 232
  Week 16 | 30.6 [22.5 to 38.8] | 60.3 [53.9 to 66.6] | 71.0 [65.1 to 77.0] | 65.5 [59.4 to 71.6]
Statistical Analysis 1: Comparison: Placebo up to Week 16 vs PF-04965842 100 mg + Placebo Injection up to Week 16; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 24.1, 95% CI 2-sided [14.0 to 34.1]
Statistical Analysis 2: Comparison: Placebo up to Week 16 vs PF-04965842 200 mg + Placebo Injection up to Week 16; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 30.1, 95% CI 2-sided [20.3 to 39.8]
Statistical Analysis 3: Comparison: Placebo up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; [analysis description as in outcome 4, analysis 3]; Test type: Other; Difference in Percentage = -2.7, 95% CI 2-sided [-9.6 to 4.2]
Statistical Analysis 4: Comparison: PF-04965842 100 mg + Placebo Injection up to Week 16 vs Dupilumab 300 mg + Oral Placebo up to Week 16; [analysis description as in outcome 4, analysis 3]; Test type: Other; Difference in Percentage = 3.1, 95% CI 2-sided [-3.3 to 9.6]

6. Secondary Outcome: Percentage of Participants Achieving EASI Response >=50% Improvement From Baseline at Week 2, 4, 8, 12 and 16
Description: EASI evaluates severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 228 | 223 | 235
  Week 2 | 21.9 [14.7 to 29.0] | 53.1 [46.6 to 59.5] | 60.5 [54.1 to 67.0] | 35.7 [29.6 to 41.9]
  Week 4: number analyzed (Participants) | 128 | 233 | 223 | 238
  Week 4 | 39.8 [31.4 to 48.3] | 73.4 [67.7 to 79.1] | 78.5 [73.1 to 83.9] | 66.8 [60.8 to 72.8]
  Week 8: number analyzed (Participants) | 129 | 232 | 224 | 239
  Week 8 | 48.8 [40.2 to 57.5] | 78.9 [73.6 to 84.1] | 88.4 [84.2 to 92.6] | 77.4 [72.1 to 82.7]
  Week 12: number analyzed (Participants) | 129 | 235 | 219 | 241
  Week 12 | 52.7 [44.1 to 61.3] | 75.3 [69.8 to 80.8] | 86.3 [81.7 to 90.9] | 80.9 [76.0 to 85.9]
  Week 16: number analyzed (Participants) | 124 | 229 | 221 | 232
  Week 16 | 57.3 [48.6 to 66.0] | 81.2 [76.2 to 86.3] | 87.3 [82.9 to 91.7] | 84.1 [79.3 to 88.8]

7. Secondary Outcome: Percentage of Participants Achieving EASI Response >=90% Improvement From Baseline at Week 2, 4, 8, 12 and 16
Description: as for outcome 6
Time Frame: Baseline, Week 2, 4, 8,12 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 228 | 223 | 235
  Week 2 | 2.3 [0.0 to 5.0] | 8.3 [4.7 to 11.9] | 11.2 [7.1 to 15.4] | 2.6 [0.5 to 4.6]
  Week 4: number analyzed (Participants) | 128 | 233 | 223 | 238
  Week 4 | 6.3 [2.1 to 10.4] | 20.2 [15.0 to 25.3] | 32.3 [26.2 to 38.4] | 12.2 [8.0 to 16.3]
  Week 8: number analyzed (Participants) | 129 | 232 | 224 | 239
  Week 8 | 7.8 [3.1 to 12.4] | 30.6 [24.7 to 36.5] | 47.3 [40.8 to 53.9] | 24.3 [18.8 to 29.7]
  Week 12: number analyzed (Participants) | 129 | 235 | 219 | 241
  Week 12 | 10.1 [4.9 to 15.3] | 36.6 [30.4 to 42.8] | 46.1 [39.5 to 52.7] | 34.9 [28.8 to 40.9]
  Week 16: number analyzed (Participants) | 124 | 229 | 221 | 232
  Week 16 | 11.3 [5.7 to 16.9] | 38.0 [31.7 to 44.3] | 48.9 [42.3 to 55.5] | 38.8 [32.5 to 45.1]

8. Secondary Outcome: Percentage of Participants Achieving EASI Response =100% Improvement From Baseline at Week 2, 4, 8, 12 and 16
Description: as for outcome 6
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 228 | 223 | 235
  Week 2 | 0 [0.0 to 2.8] | 1.3 [0.0 to 2.8] | 4.5 [1.8 to 7.2] | 0.4 [0.0 to 1.3]
  Week 4: number analyzed (Participants) | 128 | 233 | 223 | 238
  Week 4 | 0 [0.0 to 2.8] | 2.6 [0.5 to 4.6] | 7.2 [3.8 to 10.6] | 2.5 [0.5 to 4.5]
  Week 8: number analyzed (Participants) | 129 | 232 | 224 | 239
  Week 8 | 0 [0.0 to 2.8] | 6.0 [3.0 to 9.1] | 11.6 [7.4 to 15.8] | 2.1 [0.3 to 3.9]
  Week 12: number analyzed (Participants) | 129 | 235 | 219 | 241
  Week 12 | 1.6 [0.0 to 3.7] | 8.1 [4.6 to 11.6] | 12.3 [8.0 to 16.7] | 6.6 [3.5 to 9.8]
  Week 16: number analyzed (Participants) | 124 | 229 | 221 | 232
  Week 16 | 4.0 [0.6 to 7.5] | 12.7 [8.4 to 17.0] | 13.6 [9.1 to 18.1] | 5.2 [2.3 to 8.0]

9. Secondary Outcome: Time From Baseline to First Achieve at Least 4 Points Improvement in the Severity of Pruritus NRS
Description: as for outcome 3
Time Frame: Baseline up to Week 16
Population: Full analysis set till Week 16 included all randomized participants who received at least 1 dose of study medication up to Week 16. Participants with a baseline numeric rating scale score for severity of pruritus >=4 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 130 | 236 | 226 | 240
Days | NA [84.0 to NA] — Median and upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | 29.0 [16.0 to 56.0] | 13.0 [10.0 to 16.0] | 31.0 [29.0 to 57.0]

10. Secondary Outcome: Change From Baseline in Percentage Body Surface Area (BSA) at Week 2, 4, 8, 12 and 16
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: Full analysis set till Week 16 included all randomized participants who received at least 1 dose of study medication up to Week 16.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage BSA
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage BSA
  Change at Week 2 | -7.6 [-10.4 to -4.8] | -19.5 [-21.6 to -17.4] | -21.4 [-23.5 to -19.3] | -14.0 [-16.1 to -11.9]
  Change at Week 4 | -14.3 [-17.2 to -11.4] | -26.8 [-29.0 to -24.7] | -30.7 [-32.9 to -28.4] | -24.0 [-26.2 to -21.9]
  Change at Week 8 | -16.2 [-19.0 to -13.4] | -30.3 [-32.4 to -28.2] | -36.4 [-38.6 to -34.3] | -29.8 [-31.8 to -27.7]
  Change at Week 12 | -17.1 [-20.1 to -14.1] | -31.6 [-33.8 to -29.4] | -37.4 [-39.6 to -35.1] | -32.5 [-34.7 to -30.3]
  Change at Week 16 | -19.6 [-22.6 to -16.6] | -32.9 [-35.1 to -30.7] | -39.0 [-41.3 to -36.8] | -34.4 [-36.6 to -32.2]

11. Secondary Outcome: Percentage BSA at Week 18 and 20
Description: as for outcome 10
Time Frame: Week 18 and 20
Population: Full analysis set for post Week 16 included all randomized participants who received at least 1 dose of study medication post Week 16. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Percentage BSA
Groups:
- Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20: Participants who were randomized to receive oral placebo matched to PF-04965842 with subcutaneous injectable placebo matched to dupilumab till Week 16, received PF-04965842 100 mg tablet orally once daily post Week 16 up to Week 20.
- PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20: Participants who were randomized to receive PF-04965842 100 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16, received PF-04965842 100 mg tablet orally once daily post Week 16 up to Week 20.
- PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20: Participants who were randomized to receive PF-04965842 200 mg tablet orally once daily with subcutaneous injectable placebo matched to dupilumab every other week from Day 1 to Week 16, received PF-04965842 200 mg tablet orally once daily post Week 16 up to Week 20.
- Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20: Participants who were randomized to receive dupilumab 300 mg subcutaneous injection every other week with oral placebo matched to PF-04965842 once daily from Day 1 to Week 16, received oral placebo matched to PF-04965842 once daily post Week 16 up to Week 20.
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 60 | 57 | 217 | 208 | 223
Percentage BSA
  Week 18: number analyzed (Participants) | 55 | 51 | 200 | 198 | 204
  Week 18 | 22.0 (23.67) | 20.8 (22.7) | 14.8 (19.3) | 9.8 (13.6) | 13.2 (16.4)
  Week 20: number analyzed (Participants) | 57 | 56 | 212 | 197 | 214
  Week 20 | 18.0 (21.2) | 16.0 (19.7) | 14.2 (19.0) | 10.3 (14.2) | 13.2 (16.3)

12. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) at Week 2, 4, 8, 12 and 16
Description: Participant responded to the following question: "Overall, how would you describe your Atopic Dermatitis right now?" on a scale: 0= clear; 1= almost clear; 2= mild; 3= moderate; and 4= severe. Higher scores indicated more severity.
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 2 | -0.5 [-0.6 to -0.3] | -0.8 [-0.9 to -0.7] | -1.0 [-1.1 to -0.9] | -0.7 [-0.8 to -0.6]
  Change at Week 4 | -0.5 [-0.7 to -0.4] | -1.0 [-1.1 to -0.9] | -1.4 [-1.5 to -1.3] | -1.1 [-1.2 to -0.9]
  Change at Week 8 | -0.6 [-0.7 to -0.4] | -1.1 [-1.3 to -1.0] | -1.5 [-1.6 to -1.4] | -1.3 [-1.4 to -1.1]
  Change at Week 12 | -0.7 [-0.8 to -0.5] | -1.2 [-1.3 to -1.1] | -1.6 [-1.7 to -1.5] | -1.3 [-1.4 to -1.2]
  Change at Week 16 | -0.7 [-0.9 to -0.6] | -1.2 [-1.3 to -1.0] | -1.6 [-1.7 to -1.5] | -1.4 [-1.5 to -1.2]

13. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 2, 12 and 16
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Week 2, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 2 | -4.5 [-5.5 to -3.5] | -6.7 [-7.5 to -6.0] | -8.5 [-9.2 to -7.8] | -6.7 [-7.4 to -5.9]
  Change at Week 12 | -6.2 [-7.1 to -5.3] | -8.7 [-9.4 to -8.0] | -11.0 [-11.7 to -10.3] | -9.9 [-10.6 to -9.2]
  Change at Week 16 | -6.2 [-7.1 to -5.3] | -9.0 [-9.7 to -8.4] | -11.7 [-12.4 to -11.1] | -10.8 [-11.4 to -10.1]

14. Secondary Outcome: DLQI at Week 20
Description: as for outcome 13
Time Frame: Week 20
Population: Full analysis set for post Week 16 included all randomized participants who received at least 1 dose of study medication post Week 16. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 210 | 198 | 216
units on a scale | 5.3 (5.3) | 5.8 (5.7) | 6.3 (5.8) | 4.3 (4.7) | 5.6 (4.8)

15. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L) Index Value at Week 12 and 16
Description: EQ-5D-5L: standardized participant completed questionnaire consisted of 2 components: a health state profile and an optional VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprised a health state/a single utility index value. E.g. if a participant responded "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. US value sets (with all possible health states) was used for adults in the study, range from 1 to -0.109. Higher (positive) scores = better health state.
Time Frame: Baseline, Week 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 12 | 0.051 [0.032 to 0.070] | 0.101 [0.087 to 0.115] | 0.127 [0.113 to 0.141] | 0.104 [0.091 to 0.118]
  Change at Week 16 | 0.067 [0.047 to 0.087] | 0.093 [0.079 to 0.107] | 0.133 [0.119 to 0.148] | 0.113 [0.099 to 0.127]

16. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analogue Scale (VAS) Score at Week 12 and 16
Description: EQ-5D-5L consists of two components: a health state profile and an optional VAS. EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Week 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 12 | 7.975 [5.161 to 10.789] | 11.337 [9.272 to 13.401] | 17.373 [15.270 to 19.476] | 14.939 [12.900 to 16.978]
  Change at Week 16 | 7.840 [4.952 to 10.727] | 11.223 [9.129 to 13.318] | 16.711 [14.581 to 18.841] | 14.405 [12.315 to 16.496]

17. Secondary Outcome: EQ-5D-5L- Index Value at Week 20
Description: as for outcome 15
Time Frame: Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 210 | 197 | 216
units on a scale | 0.905 (0.097) | 0.894 (0.122) | 0.883 (0.124) | 0.917 (0.109) | 0.890 (0.109)

18. Secondary Outcome: EQ-5D-5L- VAS Score at Week 20
Description: as for outcome 16
Time Frame: Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 210 | 197 | 216
units on a scale | 78.2 (16.3) | 78.5 (20.2) | 76.7 (19.5) | 82.1 (17.1) | 79.6 (18.0)

19. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Anxiety Scale at Week 12 and 16
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-Anxiety (HADS-A) scale and HADS-Depression (HADS-D) scale, both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-A: sum of all 7 items resulted in score range of 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicating greater severity of anxiety.
Time Frame: Baseline, Weeks 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 12 | -0.4 [-0.9 to 0.1] | -1.2 [-1.5 to -0.8] | -1.6 [-2.0 to -1.2] | -1.4 [-1.7 to -1.0]
  Change at Week 16 | -0.4 [-0.9 to 0.1] | -1.2 [-1.6 to -0.8] | -2.0 [-2.4 to -1.6] | -1.5 [-1.9 to -1.1]

20. Secondary Outcome: Change From Baseline in HADS - Depression Scale at Week 12 and 16
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-A scale and HADS-D scale, both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-D: sum of all 7 items resulted in score range of 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicating greater severity of depression symptoms.
Time Frame: Baseline, Week 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 12 | -0.3 [-0.7 to 0.2] | -1.3 [-1.6 to -0.9] | -1.6 [-1.9 to -1.2] | -1.3 [-1.6 to -0.9]
  Change at Week 16 | -0.3 [-0.8 to 0.2] | -1.0 [-1.4 to -0.7] | -1.6 [-1.9 to -1.2] | -1.2 [-1.5 to -0.8]

21. Secondary Outcome: HADS - Anxiety Scale at Week 20
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-A scale and HADS-D scale, both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-A: sum of all 7 items resulted in score range of 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicating greater severity of anxiety.
Time Frame: Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 209 | 197 | 215
units on a scale | 3.4 (3.2) | 4.5 (4.5) | 4.0 (3.8) | 3.1 (3.1) | 3.7 (3.5)

22. Secondary Outcome: HADS - Depression Scale at Week 20
Description: as for outcome 20
Time Frame: Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 209 | 197 | 215
units on a scale | 2.6 (3.4) | 3.6 (3.7) | 2.8 (3.2) | 2.2 (3.1) | 2.7 (3.3)

23. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) at Week 12 and 16
Description: POEM is a 7-item participant reported outcome (PRO) measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item is scored as following: "no days (0)", "1-2 days (1)", "3-4 days (2)", "5-6 days (3)" and "every day (4)". The score ranges from 0 to 28, where higher score indicated greater severity.
Time Frame: Baseline, Week 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 241
units on a scale
  Change at Week 12 | -5.1 [-6.3 to -3.9] | -9.6 [-10.5 to -8.6] | -12.6 [-13.6 to -11.7] | -10.8 [-11.7 to -9.9]
  Change at Week 16 | -5.0 [-6.3 to -3.8] | -9.2 [-10.1 to -8.2] | -12.5 [-13.4 to -11.6] | -10.8 [-11.8 to -9.9]

24. Secondary Outcome: POEM at Week 20
Description: as for outcome 23
Time Frame: Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 55 | 55 | 209 | 196 | 215
units on a scale | 10.7 (6.8) | 9.6 (7.8) | 11.6 (7.7) | 8.6 (7.0) | 11.0 (6.9)

25. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis (PSAAD) Total Score Week 1 to Week 16
Description: PSAAD is a daily participant reported symptom electronic diary. Participants rated their symptoms of AD over the past 24 hours, using 11 items (itchy skin, painful skin, dry skin, flaky skin, cracked skin, bumpy skin, red skin, discolored skin [lighter or darker], bleeding from skin, seeping or oozing fluid from skin [other than blood], and skin swelling). Participant had to think about all the areas of their body affected by their skin condition and chose the number that best described their experience for each of the 11 items, from 0 (no symptoms) to 10 (extreme symptoms), higher scores signified worse skin condition. Total PSAAD score = arithmetic mean of 11 items, 0 (no symptoms) to 10 (extreme symptoms), where higher score = worse skin condition.
Time Frame: Baseline, Week 1 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 130 | 237 | 225 | 241
units on a scale
  Change at Week 1 | -0.5 [-0.8 to -0.3] | -1.1 [-1.3 to -0.9] | -1.3 [-1.5 to -1.2] | -0.9 [-1.1 to -0.8]
  Change at Week 2 | -0.9 [-1.2 to -0.7] | -1.8 [-2.0 to -1.6] | -2.3 [-2.5 to -2.1] | -1.6 [-1.8 to -1.4]
  Change at Week 3 | -1.1 [-1.4 to -0.8] | -2.2 [-2.4 to -2.0] | -2.8 [-3.0 to -2.6] | -2.1 [-2.3 to -1.9]
  Change at Week 4 | -1.4 [-1.7 to -1.1] | -2.4 [-2.6 to -2.2] | -3.0 [-3.3 to -2.8] | -2.4 [-2.7 to -2.2]
  Change at Week 5 | -1.5 [-1.8 to -1.2] | -2.6 [-2.8 to -2.4] | -3.2 [-3.5 to -3.0] | -2.7 [-2.9 to -2.5]
  Change at Week 6 | -1.5 [-1.8 to -1.2] | -2.6 [-2.8 to -2.4] | -3.3 [-3.6 to -3.1] | -2.8 [-3.1 to -2.6]
  Change at Week 7 | -1.6 [-1.9 to -1.2] | -2.7 [-2.9 to -2.4] | -3.4 [-3.6 to -3.1] | -2.9 [-3.2 to -2.7]
  Change at Week 8 | -1.5 [-1.9 to -1.2] | -2.7 [-2.9 to -2.4] | -3.4 [-3.7 to -3.2] | -3.0 [-3.2 to -2.7]
  Change at Week 9 | -1.7 [-2.0 to -1.4] | -2.7 [-2.9 to -2.4] | -3.5 [-3.8 to -3.3] | -3.1 [-3.3 to -2.8]
  Change at Week 10 | -1.7 [-2.0 to -1.4] | -2.7 [-2.9 to -2.4] | -3.5 [-3.8 to -3.3] | -3.1 [-3.4 to -2.9]
  Change at Week 11 | -1.6 [-1.9 to -1.3] | -2.7 [-2.9 to -2.4] | -3.5 [-3.8 to -3.3] | -3.2 [-3.4 to -2.9]
  Change at Week 12 | -1.6 [-2.0 to -1.3] | -2.7 [-3.0 to -2.5] | -3.6 [-3.8 to -3.3] | -3.2 [-3.5 to -3.0]
  Change at Week 13 | -1.7 [-2.0 to -1.4] | -2.8 [-3.1 to -2.6] | -3.7 [-3.9 to -3.4] | -3.3 [-3.6 to -3.1]
  Change at Week 14 | -1.6 [-1.9 to -1.3] | -2.8 [-3.1 to -2.6] | -3.6 [-3.9 to -3.4] | -3.4 [-3.6 to -3.2]
  Change at Week 15 | -1.7 [-2.0 to -1.4] | -2.9 [-3.1 to -2.6] | -3.6 [-3.8 to -3.4] | -3.4 [-3.6 to -3.1]
  Change at Week 16 | -1.7 [-2.0 to -1.3] | -2.8 [-3.1 to -2.6] | -3.6 [-3.8 to -3.4] | -3.4 [-3.6 to -3.2]

26. Secondary Outcome: PSAAD Total Score at Week 18 and 20
Description: as for outcome 25
Time Frame: Week 18 and 20
Population: Full analysis set for post Week 16 included all randomized participants who received at least 1 dose of study medication post Week 16. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 54 | 54 | 202 | 202 | 218
units on a scale
  Week 18 | 2.6 (1.9) | 3.0 (2.4) | 2.2 (1.9) | 1.7 (1.7) | 1.8 (1.5)
  Week 20: number analyzed (Participants) | 54 | 53 | 201 | 199 | 213
  Week 20 | 2.5 (2.0) | 2.6 (2.3) | 2.2 (1.9) | 1.8 (1.8) | 2.0 (1.6)

27. Secondary Outcome: Percentage of Participants With Scoring Atopic Dermatitis (SCORAD) Response >=50% Improvement From Baseline at Week 2, 4, 8, 12 and 16
Description: SCORAD: scoring index for AD combining extent, severity, subjective symptoms. Extent (A): rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none=0, mild=1, moderate=2,severe=3. The severity scores were summed to give B (0-18). Subjective symptoms (C): pruritus and sleep, each of these 2 were scored by participant/caregiver using visual analogue scale (VAS) where "0" = no itch/no sleeplessness and "10" = the worst imaginable itch/sleeplessness, higher scores=worse symptoms. Scores for itch and sleeplessness were added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD=worse outcome.
Time Frame: Baseline, Week 2, 4, 8 12 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 233 | 224 | 237
  Week 2 | 10.2 [4.9 to 15.4] | 23.6 [18.2 to 29.1] | 38.4 [32.0 to 44.8] | 15.6 [11.0 to 20.2]
  Week 4: number analyzed (Participants) | 129 | 234 | 224 | 238
  Week 4 | 18.6 [11.9 to 25.3] | 45.7 [39.3 to 52.1] | 61.6 [55.2 to 68.0] | 45.8 [39.5 to 52.1]
  Week 8: number analyzed (Participants) | 129 | 234 | 225 | 239
  Week 8 | 20.2 [13.2 to 27.1] | 53.4 [47.0 to 59.8] | 71.6 [65.7 to 77.5] | 56.9 [50.6 to 63.2]
  Week 12: number analyzed (Participants) | 128 | 234 | 224 | 238
  Week 12 | 27.3 [19.6 to 35.1] | 56.8 [50.5 to 63.2] | 72.3 [66.5 to 78.2] | 64.3 [58.2 to 70.4]
  Week 16: number analyzed (Participants) | 123 | 228 | 221 | 231
  Week 16 | 33.3 [25.0 to 41.7] | 56.1 [49.7 to 62.6] | 68.8 [62.7 to 74.9] | 67.5 [61.5 to 73.6]

28. Secondary Outcome: Percentage of Participants With SCORAD Response >=75% Improvement From Baseline at Week 2, 4, 8 12 and 16
Description: as for outcome 27
Time Frame: Baseline, Week 2, 4, 8 12 and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Percentage of participants
  Week 2: number analyzed (Participants) | 128 | 233 | 224 | 237
  Week 2 | 1.6 [0.0 to 3.7] | 6.4 [3.3 to 9.6] | 8.5 [4.8 to 12.1] | 0.8 [0.0 to 2.0]
  Week 4: number analyzed (Participants) | 129 | 234 | 224 | 238
  Week 4 | 3.1 [0.1 to 6.1] | 12.4 [8.2 to 16.6] | 25.4 [19.7 to 31.2] | 7.1 [3.9 to 10.4]
  Week 8: number analyzed (Participants) | 129 | 234 | 225 | 239
  Week 8 | 3.1 [0.1 to 6.1] | 19.2 [14.2 to 24.3] | 41.3 [34.9 to 47.8] | 16.3 [11.6 to 21.0]
  Week 12: number analyzed (Participants) | 128 | 234 | 224 | 238
  Week 12 | 6.3 [2.1 to 10.4] | 25.6 [20.0 to 31.2] | 39.3 [32.9 to 45.7] | 26.1 [20.5 to 31.6]
  Week 16: number analyzed (Participants) | 123 | 228 | 221 | 231
  Week 16 | 10.6 [5.1 to 16.0] | 26.8 [21.0 to 32.5] | 40.3 [33.8 to 46.7] | 29.4 [23.6 to 35.3]

29. Secondary Outcome: Change From Baseline in SCORAD Visual Analogue Scale (VAS) of Itch and Sleep Loss at Week 2, 4, 8 12 and 16
Description: as for outcome 27
Time Frame: Baseline, Week 2, 4, 8 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 129 | 237 | 225 | 241
units on a scale
  Itch: Change at Week 2 | -1.5 [-1.9 to -1.2] | -2.9 [-3.2 to -2.7] | -3.7 [-4.0 to -3.4] | -2.4 [-2.7 to -2.1]
  Itch: Change at Week 4 | -2.2 [-2.6 to -1.8] | -3.7 [-4.0 to -3.4] | -4.6 [-4.9 to -4.3] | -3.7 [-4.0 to -3.4]
  Itch: Change at Week 8 | -2.3 [-2.7 to -1.9] | -3.9 [-4.2 to -3.6] | -4.9 [-5.2 to -4.6] | -4.2 [-4.5 to -3.9]
  Itch: Change at Week 12 | -2.4 [-2.9 to -2.0] | -3.9 [-4.3 to -3.6] | -5.0 [-5.3 to -4.7] | -4.4 [-4.7 to -4.1]
  Itch: Change at Week 16 | -2.7 [-3.1 to -2.3] | -3.8 [-4.1 to -3.5] | -4.8 [-5.1 to -4.5] | -4.5 [-4.8 to -4.2]
  Sleep loss: Change at Week 2 | -1.6 [-2.0 to -1.2] | -2.6 [-2.9 to -2.3] | -3.3 [-3.6 to -3.0] | -2.3 [-2.6 to -1.9]
  Sleep loss: Change at Week 4 | -2.3 [-2.7 to -1.9] | -3.4 [-3.7 to -3.1] | -4.2 [-4.5 to -3.9] | -3.4 [-3.7 to -3.1]
  Sleep loss: Change at Week 8 | -2.3 [-2.7 to -1.9] | -3.6 [-3.9 to -3.3] | -4.4 [-4.7 to -4.1] | -3.9 [-4.2 to -3.6]
  Sleep loss: Change at Week 12 | -2.4 [-2.8 to -2.0] | -3.7 [-4.0 to -3.4] | -4.6 [-4.9 to -4.3] | -4.2 [-4.5 to -3.9]
  Sleep loss: Change at Week 16 | -2.6 [-3.0 to -2.2] | -3.7 [-4.0 to -3.4] | -4.8 [-5.1 to -4.5] | -4.3 [-4.6 to -4.0]

30. Secondary Outcome: SCORAD VAS of Itch and Sleep Loss at Week 18 and 20
Description: as for outcome 27
Time Frame: Week 18 and 20
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
Number analyzed (Participants) | 60 | 57 | 217 | 208 | 223
units on a scale
  Itch: Week 18: number analyzed (Participants) | 56 | 52 | 204 | 201 | 206
  Itch: Week 18 | 3.2 (2.6) | 2.7 (2.2) | 3.0 (2.5) | 2.3 (2.2) | 2.7 (2.2)
  Itch: Week 20: number analyzed (Participants) | 58 | 57 | 212 | 199 | 218
  Itch: Week 20 | 2.9 (2.4) | 2.6 (2.4) | 3.2 (2.6) | 2.3 (2.3) | 2.8 (2.2)
  Sleep loss: Week 18: number analyzed (Participants) | 56 | 52 | 204 | 201 | 206
  Sleep loss: Week 18 | 2.2 (2.3) | 2.3 (2.3) | 2.1 (2.3) | 1.6 (2.1) | 1.8 (2.0)
  Sleep loss: Week 20: number analyzed (Participants) | 58 | 57 | 212 | 199 | 218
  Sleep loss: Week 20 | 2.1 (2.2) | 2.0 (2.3) | 2.4 (2.6) | 1.5 (2.1) | 1.7 (2.1)

31. Secondary Outcome: Least Square Mean of Number of Steroid-free Days From Baseline up to Week 16
Description: Number of days when a corticosteroid as a concomitant medication was not used up to Week 16 is reported as Least square mean in this outcome measure.
Time Frame: Baseline up to Week 16
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16
Number analyzed (Participants) | 131 | 238 | 226 | 242
Days | 21.8 [14.9 to 28.8] | 30.2 [25.1 to 35.4] | 33.6 [28.3 to 38.9] | 28.1 [23.0 to 33.2]

ADVERSE EVENTS:
Time Frame: For reporting arms till Week 16 analysis: Baseline up to Week 16; For reporting arms post Week 16 analysis: Week 16 to Week 24 (28 days after last dose of study drug)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Placebo up to Week 16 | PF-04965842 100 mg + Placebo Injection up to Week 16 | PF-04965842 200 mg + Placebo Injection up to Week 16 | Dupilumab 300 mg + Oral Placebo up to Week 16 | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/238 | 0/226 | 0/242 | 0/60 | 0/57 | 0/217 | 0/208 | 0/223
Serious Adverse Events (participants affected / at risk) | 5/131 | 6/238 | 2/226 | 2/242 | 0/60 | 0/57 | 1/217 | 0/208 | 1/223
Other Adverse Events (participants affected / at risk) | 68/131 | 121/238 | 140/226 | 120/242 | 13/60 | 16/57 | 50/217 | 45/208 | 31/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo up to Week 16 (N=131) | PF-04965842 100 mg + Placebo Injection up to Week 16 (N=238) | PF-04965842 200 mg + Placebo Injection up to Week 16 (N=226) | Dupilumab 300 mg + Oral Placebo up to Week 16 (N=242) | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 (N=60) | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 (N=57) | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 (N=217) | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 (N=208) | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20 (N=223)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo up to Week 16 (N=131) | PF-04965842 100 mg + Placebo Injection up to Week 16 (N=238) | PF-04965842 200 mg + Placebo Injection up to Week 16 (N=226) | Dupilumab 300 mg + Oral Placebo up to Week 16 (N=242) | Placebo up to Week 16 Then PF-04965842 100 mg Week 16 to 20 (N=60) | Placebo up to Week 16 Then PF-04965842 200 mg Week 16 to 20 (N=57) | PF-04965842 100 mg + Placebo Injection up to Week 16 Then PF-04965842 100 mg Week 16 to 20 (N=217) | PF-04965842 200 mg + Placebo Injection up to Week 16 Then PF-04965842 200 mg Week 16 to 20 (N=208) | Dupilumab 300 mg + Oral Placebo up to Week 16 Then Oral Placebo Week 16 to 20 (N=223)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Defect conduction intraventricular (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Congenital lacrimal passage anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Conjunctival irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dry eye (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eye irritation (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eye pain (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eye pruritus (Eye disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eyelid oedema (Eye disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eyelid pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Noninfective conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Presbyopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eczema eyelids (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eyelid cyst (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dental caries (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 4 | 3 | 0 | 2 | 3 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nausea (Gastrointestinal disorders) | 2 | 10 | 25 | 7 | 0 | 5 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 4 | 0 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Asthenia (General disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Chest pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Fatigue (General disorders) | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Injection site oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Injection site pain (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Medical device site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Oedema peripheral (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pyrexia (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Swelling (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Swelling face (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Therapeutic response unexpected (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Xerosis (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Allergy to chemicals (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Abscess limb (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Body tinea (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Cellulitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Conjunctivitis (Infections and infestations) | 3 | 2 | 3 | 15 | 0 | 0 | 0 | 0 | 2 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eczema herpeticum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Folliculitis (Infections and infestations) | 4 | 4 | 4 | 2 | 0 | 1 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Furuncle (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Herpes simplex (Infections and infestations) | 1 | 5 | 8 | 2 | 0 | 0 | 1 | 4 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Herpes zoster (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hordeolum (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Impetigo (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Kaposi's varicelliform eruption (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Malassezia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nasopharyngitis (Infections and infestations) | 9 | 22 | 15 | 23 | 3 | 2 | 3 | 9 | 5 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Oral herpes (Infections and infestations) | 1 | 3 | 2 | 5 | 0 | 1 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Paronychia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Perichondritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pharyngitis (Infections and infestations) | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pulpitis dental (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pustule (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 3 | 0 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin candida (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tinea versicolour (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Upper respiratory tract infection (Infections and infestations) | 6 | 12 | 9 | 9 | 1 | 0 | 6 | 5 | 7 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ureaplasma infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urinary tract infection (Infections and infestations) | 2 | 4 | 7 | 4 | 2 | 0 | 2 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nasal herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Medication error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Biopsy endometrium (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood creatine phosphokinase increased (Investigations) | 3 | 7 | 6 | 2 | 1 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Electrocardiogram T wave amplitude increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Haemoglobin decreased (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Lipids increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Natural killer cell count decreased (Investigations) | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Red blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
T-lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 7 | 0 | 0 | 1 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Mandibular mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dizziness (Nervous system disorders) | 2 | 4 | 7 | 0 | 0 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
External compression headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Headache (Nervous system disorders) | 6 | 10 | 15 | 13 | 1 | 1 | 2 | 0 | 2 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypertonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Somnolence (Nervous system disorders) | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Apathy (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urinary tract inflammation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ovarian disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 3 | 0 | 0 | 3 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Acne (Skin and subcutaneous tissue disorders) | 0 | 7 | 15 | 3 | 1 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 7 | 3 | 2 | 0 | 0 | 1 | 4 | 2 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Victim of crime (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Rotator cuff repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Essential hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Hypertension (Vascular disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 1 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.
Eosinophil percentage increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v22.1 was used for coding events till Week 16 and MedDRA v23.0 was used for coding events post Week 16.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03720470/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03720470/SAP_001.pdf